CLINICAL TRIAL: NCT06501521
Title: Non-invasive Brain Tumor Diagnosis Through Analysis of Proximal Fluids, Circulating Tumor Cells, and Biomolecules
Brief Title: Non-invasive Brain Tumor Molecular Diagnostics and Monitoring
Status: Recruiting | Type: Observational
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: NW25-03-00198
Record Dates: First submitted 2024-07-01; First posted 2024-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. ocular secretion
  2. peripheral blood
  3. urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Glioblastoma multiforme: Patients with GBM
  Interventions: Diagnostic Test: Diagnostic test
- Low-grade glioma: Patients with low-grade gliomas.
  Interventions: Diagnostic Test: Diagnostic test
- Control group: Patients without cancer or systemic inflammation
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — No intervention among the arms. The diagnostic, prognostic, predictive and follow-up value of tested biomolecules will be analyzed.

SUMMARY:
This prospective multicenter study aims to enroll GBM patients who will undergo repeated assessments (preoperatively and 3 months post-surgery) to detect circulating tumor cells and analyze the transcriptomic profiles of EVs in their blood. The prognostic and monitoring significance of these biomarkers to disease course (assessing treatment efficacy, resistance incidence, tumor progression) will be evaluated.

Concurrently, proteomic profiles typical of GBM will be analyzed in blood and ocular secretion samples from GBM patients, patients with low-grade gliomas, and patients without brain tumors to identify and validate novel protein biomarkers suitable for disease monitoring. Additionally, this study proposes an innovative approach to monitor GBM patients by investigating the presence of GBM-specific nucleic acid fragments in urine.

ELIGIBILITY:
Inclusion Criteria: Adult patients with brain tumors -

Exclusion Criteria: No other cancer; no inflammatory disease

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inhabitants of Olomouc region
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Proteomic profiles of proximal liquids in brain tumor patients | 2020-2023
  The protein profiles will be measured in ocular secretion and plasma samples of patients wiht GBM, low-grade glioma and control cohort. Candidate proteins will be correleted with clinical parameters. The number of patients with identified prognostic biomarkers will be reported.
Circulating tumor cells (CTCs) for non-invasive monitoring of GBM patients. | 2020-2030
  The number of CTCs and their molecular characteristics will be measured in peripheral blod of GBM patients. The CTCs counts will be correleted with the clinical parameters. The number of patients with the presence or absence of CTCs will be reported.
Extracellular vesicles (EVs) for non-invasive monitoring of GBM patients. | 2020-2030
  The RNA profiles of EVs will be measured in plasma samples of patients wiht GBM. Candidate RNAs will be correleted with clinical parameters. The number of patients with identified prognostic RNAs will be reported.
Urine as a source of GBM-specific nucleic acids fragments for disease monitoring. | 2025-2030
  The GBM-specific nucleic acids fragments will be measured in urine of GBM patients. Candidate nucleic acids will be correleted with clinical parameters. The number of patients with identified prognostic biomolecules will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD,PhD, Principal Investigator — Faculty of Medicine and Dentistry, Palacky University Olomouc, Czech Republic
Locations (1):
- Department of Neurosurgery, University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous proteomic profiles of plasma and ocular secretion and transcriptomic data from extracelular vesicles will be shared.